CLINICAL TRIAL: NCT04796194
Title: A Phase 2 Study of Intratumoral Injection of LTX-315 in Combination With Pembrolizumab in Patients With Percutaneously Accessible Lesions With Advanced Melanoma Refractory to PD-1/PD-L1 Inhibitor Therapy.
Brief Title: Intratumoral Injection of LTX-315 in Combination With Pembrolizumab in Advanced Melanoma
Acronym: ATLAS-IT-05
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lytix Biopharma AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C20-315-05 (ATLAS-IT-05)
Record Dates: First submitted 2021-03-02; First posted 2021-03-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Advanced Melanoma
Keywords: Oncolytic peptide; LTX-315; Pembrolizumab; Intratumoral; Melanoma
MeSH Terms: conditions — Melanoma | interventions — LTX-315; pembrolizumab

STUDY DESIGN:
Intervention Model Description: LTX-315 in Combination With Pembrolizumab
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LTX-315 in combination with pembrolizumab (Experimental): LTX-315 will be injected directly into the selected tumor lesion(s).
  Pembrolizumab will be dispensed and administered as an IV infusion.
  Interventions: Combination Product: LTX-315 in combination with pembrolizumab

INTERVENTIONS:
Combination Product: LTX-315 in combination with pembrolizumab — Phase A Pembrolizumab will be given as 200 mg IV infusion over 30 minutes on Days 1 and 22.
  Phase B Pembrolizumab will be given as 400 mg IV infusion over 30 minutes every 6 weeks starting at Day 43 (3 weeks after the last dose of pembrolizumab in Phase A) until discontinuation from the study or for a maximum of 24 months' total therapy, whichever comes first.

SUMMARY:
ATLAS-IT-05 is an open-label, single-arm study in patients with advanced melanoma accessible for injections (cutaneous, subcutaneous, lymph node, or intramuscular tumors) and who have either exhausted treatment options or are not eligible for, suitable for, or willing to undergo such treatments.

DETAILED DESCRIPTION:
The study aims to assess the safety and efficacy of LTX-315 in combination with the immune checkpoint inhibitor (ICI) pembrolizumab in patients with advanced melanoma.

LTX-315 has been administered with pembrolizumab in a previous Phase I/II study, and there were clear indications that LTX-315 + pembrolizumab was a clinically active combination. Furthermore, the addition of LTX-315 to pembrolizumab dosing did not appear to increase the overall incidence or severity profile of toxicities.

The present study will document the preliminary efficacy, clinical safety, and tolerability of LTX-315 in combination with pembrolizumab, in a dose and regimen that is considered to be safe.

Patient population consists of patients with stage III B, C, D and Stage IVm1a, m1b unresectable metastatic melanoma with ECOG performance status of 0 or 1, who have received an FDA-approved anti-PD/PD-L1 therapy and have progressed after prior anti-PD-1 or anti-PD-L1 therapy, alone or in combination with systemic therapy.

ELIGIBILITY:
The following are the main INCLUSION CRITERIA:

Diagnosis and main criteria for inclusion and exclusion:

The following are the main inclusion criteria:

1. Have one of the following confirmed histologically:

   Patients with Stage III B, C, D or Stage IV m1a, m1b unresectable metastatic melanoma who have received an approved anti-PD-1/PD-L1 therapy and have progressed on or after prior anti-PD-1 or anti-PD-L1 therapy, alone or in combination with systemic therapy.

   For patients who have refused prior standard-of-care treatment other than anti-PD-1/PDL-1 therapy, the patient's reason for refusing standard therapy for their disease shall be clearly documented in the study electronic case report form prior to study participation.

   All patients must have received anti-PD-1 or anti-PD-L1 in addition to complying with the relevant criteria below. Melanoma patients with v-raf murine sarcoma viral oncogene homolog B1 (BRAF) mutation who are eligible and suitable for BRAF inhibitor therapy should have received specific BRAF inhibitor therapy before enrolling in this study and must have completed treatments at least 3 weeks prior to starting treatment and have no signs of rapidly progressive disease (PD). Patients who have refused BRAF inhibitor therapy are also eligible for the study.
2. The patients should have had radiologically PD after the most recent line of systemic therapy (no more than two prior lines in the metastatic setting). Adjuvant or Neoadjuvant therapy is not considered as a prior line of treatment for eligibility purposes. Anti-PD-1 or anti-PD-L1 does not need to be the most recent line of therapy prior to study entry.
3. Disease that is not amenable to further radiotherapy or surgery for cancer treatment.
4. Have at least one superficial, non-visceral tumor lesion accessible for injection via cutaneous, subcutaneous, or intramuscular route. Note, lymph nodes with metastatic disease may be selected for injection if they are superficial, but not if deep-seated; visceral lesions must not be selected for injection. The lesion must not be located close to airways, defined as close enough to jeopardize the patient's safety, in the opinion of the Investigator, in the event of a local reaction to LTX-315 injection (for example, if such a reaction has the potential to interfere with swallowing or result in hemorrhaging into the airways). The size of the lesion(s) selected for injection must be ≤2 cm in the mean longest perpendicular diameter. For larger lesions or conglomerate lesions, approval from the sponsor's Medical Monitor is needed prior to enrollment.
5. At least one measurable target lesion evaluable according to RECIST version 1.1 that is not planned to be injected with LTX-315 or biopsied. The location of this noninjected tumor may be superficial, deep-seated, or visceral.
6. Have a life expectancy ≥3 months.
7. Are males or females aged 18 years or older.
8. Have an ECOG performance status of 0 or 1.
9. Resolution of all disease or prior treatment-related toxicities to Grade ≤1, with the exception of alopecia, <Grade 2 neuropathy and laboratory abnormalities (parameters below apply). If the patient underwent major surgery or received radiation therapy, they must have fully recovered from the intervention.
10. Have a left ventricular ejection fraction (LVEF) that is above the institution's lower limit of normal (by echo scan assessment).
11. Meet the following laboratory requirements:

    1. Absolute neutrophil count ≥1.00 × 109/L,
    2. Absolute lymphocyte count that is ≥0.5 k/µL or equivalent,
    3. Platelet count ≥75.0 × 109/L,
    4. Hemoglobin ≥9.0 g/dL,
    5. Prothrombin time/partial thromboplastin time ≤1.5 x upper limit of normal (ULN), if the patient is receiving oral anticoagulation international normalized ratio ≤1.5 x ULN, activated partial thromboplastin time ≤1.5 x ULN,
    6. Total bilirubin ≤1.5 x ULN (≤2 x ULN if associated with hepatobiliary metastases or Gilbert's syndrome) AND associated to the aspartate aminotransferase (AST) and alanine aminotransferase (ALT) 2.5 x ULN,
    7. AST and ALT ≤2.5 × ULN,
    8. Calculated creatinine clearance ≥30 mL/min using Cockcroft-Gault formula,
    9. Lactate dehydrogenase (LDH) ≤ULN,
    10. Serum albumin ≥30g/L.
12. Are willing and able to comply with the protocol and agree to return to the clinical site for follow-up visits and examinations.
13. Are willing to undergo tumor biopsy procedures.
14. Are fully informed about the study and have signed the informed consent form (ICF).
15. Are willing to use contraceptive measures as prescribed by the protocol. Female patients of childbearing potential and their partners who are sexually active must agree to the use of two highly effective forms of contraception starting from the screening visit, throughout their participation in the study, and for at least 120 days after their last dose of pembrolizumab or at least 180 days after their last dose of LTX-315, whichever is longer. Male patients with partners who are pregnant or of childbearing potential must use a barrier method of contraception starting from the screening visit, throughout their participation in the study and for at least 120 days after their last dose of pembrolizumab or at least 180 days after their last dose of LTX 315, whichever is longer. A woman is considered of childbearing potential, that is, fertile, following menarche and until becoming postmenopausal unless permanently sterile.
16. Female patients must not be pregnant or breastfeeding. Female patients of childbearing potential must have a negative pregnancy test result during screening and at Day 1.

The following are the main exclusion criteria:

1. Patients with primary ocular melanoma or mucosal melanoma are not eligible
2. Has excessive tumor burden. The patient has more than 10 lesions available for injection, or has any injected lesion >2cm, or in the opinion of the Investigator. For larger lesions or conglomerate lesions, approval from the sponsor's Medical Monitor is needed prior to enrollment. Patients with more than 10 lesions may be deemed eligible after discussion with the sponsor's Medical Monitor, based on assessment of overall tumor burden.
3. Known bone-only or active central nervous system metastases and/or carcinomatous meningitis.

   Patients with untreated brain metastases ≤3 mm that are asymptomatic, do not have significant edema, and do not require steroids or anti-seizure medications are eligible after discussion with the sponsor's Medical Monitor. Patients with previously treated brain metastases may participate provided they are stable after treatment and without evidence of progression by imaging for at least 4 weeks prior to the first dose of study drug administration, and are not using corticosteroids for at least 7 days prior to study drug administration.
4. Have a history of cerebrovascular or cardiac disorders (e.g., Class III or IV New York Heart Association cardiac failure) and in the investigators' opinion the patient would be at particular risk of sequelae following a short hypotensive episode.
5. Have a marked baseline prolongation of QT interval corrected for heart rate using Fridericia's formula (i.e., repeated demonstration of a QTc interval >480 ms National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] Grade 2).
6. Are currently taking immunosuppressive agents or use of systemic corticosteroids or other systemic immunosuppressive drugs within 28 days prior to study drug administration (see Appendix 4 for examples). Patients who require corticosteroids should have been on a stable dose (up to 10 mg daily prednisone or equivalent) for at least 2 weeks prior to study drug administration. Topical and inhaled corticosteroids are also permitted.
7. Have a history of systemic autoimmune disease requiring anti-inflammatory or immunosuppressive therapy within 3 months prior to Day 1, with the following exceptions:

   1. Patients with a history of autoimmune thyroiditis are eligible provided they require only thyroid hormone replacement therapy and their disease has been stable for ≥1 year.
   2. Patients with well-controlled type I diabetes (in the opinion of the Investigator) are eligible.
   3. Patients with a history of chronic disease, who have been stable for the preceding 6 months without treatment.
8. Patients who are allergic or have hypersensitivity to chlorpheniramine or equivalent H1 antagonist, cimetidine or equivalent H2 antagonist, or montelukast.
9. Have a history of severe hypersensitivity to another monoclonal antibody; are receiving immunosuppressive therapy; have a history of severe immune-related adverse reaction from treatment with a monoclonal antibody, defined as any Grade ≥3 toxicity requiring corticosteroid treatment (>10 mg/day prednisone or equivalent) for >12 weeks.
10. Have had (non-infectious) pneumonitis Grade ≥3 in the past or current pneumonitis.
11. History of interstitial lung disease.
12. Have a known hypersensitivity to pembrolizumab or LTX-315 or any of their excipients (for pembrolizumab those listed in the prescribing information).
13. Have any other serious illness or medical condition, such as, but not limited to:

    1. Uncontrolled infection or infection requiring systemic antibiotics,
    2. Uncontrolled cardiac failure: Class III or IV New York Heart Association,
    3. Uncontrolled hypertension or risk factors for uncontrolled hypertension (>160 mmHg systolic and/or >100 mmHg diastolic), despite appropriate antihypertensive medication,
    4. Uncontrolled systemic or gastrointestinal inflammatory conditions,
    5. Known bone marrow dysplasia,
    6. History of positive tests for human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome or active hepatitis B or C (based on serology); positive serology will be confirmed by a viral load test. Patients with treated HIV and a viral load test result consistent with treated HIV, as well as patients with treated hepatitis B or C with an undetectable viral load test result, are eligible,
    7. History of or current mastocytosis.
14. Have received external radiotherapy or cytotoxic chemotherapy within 4 weeks prior to Day 1 or have not recovered (to NCI-CTCAE Grade ≤1; alopecia of any grade is allowed, and peripheral neuropathy of up to Grade 2 is allowed) from adverse events (AEs) due to such agents being administered more than 4 weeks prior to Day 1.
15. Have received cancer immunotherapy within 4 weeks prior to Day 1 or have not recovered from AEs (to NCI-CTCAE Grade ≤1) due to such agents being administered more than 4 weeks prior to Day 1.
16. Have received an investigational drug within 4 weeks prior to Day 1 or are scheduled to receive one during the treatment or post-treatment periods.
17. Are expected to need any other anticancer therapy or immunotherapy to be initiated during the study period. Note: Palliative radiotherapy or surgery are allowable under certain conditions in Phase B.
18. Receipt of any BRAF and/or mitogen-activated protein kinase (MEK) inhibitor (including any investigational inhibitor) within 3 weeks before first dose of study drug and/or with signs of rapidly progressive disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Through study completion, an average of 6 months
  ...defined as the proportion of patients who achieved partial response (PR) and/or complete response (CR) per local investigator assessment using RECIST version 1.1.
Clinical benefit rate (CBR) | Through study completion, an average of 6 months
  ...defined as the proportion of patients who respond to treatment, estimated as the proportion of patients who achieve stable disease (SD), PR, or CR per local investigator assessment using RECIST version 1.1
Overall survival (OS) | Through study completion, an average of 6 months
  ...evaluated as time from baseline until death

CONTACTS AND LOCATIONS:
Overall Officials: Oystein Rekdal, PHD, Study Director — Lytix Biopharma
Locations (10):
- United States (4):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Levine Cancer Institute - Atrium Health, Charlotte, North Carolina
  - University of Pittsburgh Medical Center (UPMC) Hilman Cancer Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Centre, Houston, Texas
- France (3):
  - Centre Hospitalier Regional Universitaire De Lille, Lille
  - Gustave Roussy Cancer Campus, Paris
  - Hospital Lyon Sud, Pierre-Bénite
- Norway (2):
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital--Radiumhospitalet, Oslo
- Clínica Universidad de Navarra, Pamplona, Spain

REFERENCES:
- [Background] Camilio KA, Rekdal O, Sveinbjornsson B. LTX-315 (Oncopore): A short synthetic anticancer peptide and novel immunotherapeutic agent. Oncoimmunology. 2014 Jun 25;3:e29181. doi: 10.4161/onci.29181. eCollection 2014. PMID 25083333
- [Background] Sveinbjornsson B, Camilio KA, Haug BE, Rekdal O. LTX-315: a first-in-class oncolytic peptide that reprograms the tumor microenvironment. Future Med Chem. 2017 Aug;9(12):1339-1344. doi: 10.4155/fmc-2017-0088. Epub 2017 May 11. PMID 28490192
- [Background] Jebsen NL, Apelseth TO, Haugland HK, Rekdal O, Patel H, Gjertsen BT, Jossang DE. Enhanced T-lymphocyte infiltration in a desmoid tumor of the thoracic wall in a young woman treated with intratumoral injections of the oncolytic peptide LTX-315: a case report. J Med Case Rep. 2019 Jun 10;13(1):177. doi: 10.1186/s13256-019-2088-6. PMID 31177991
- [Background] Spicer J, Marabelle A, Baurain JF, Jebsen NL, Jossang DE, Awada A, Kristeleit R, Loirat D, Lazaridis G, Jungels C, Brunsvig P, Nicolaisen B, Saunders A, Patel H, Galon J, Hermitte F, Camilio KA, Mauseth B, Sundvold V, Sveinbjornsson B, Rekdal O. Safety, Antitumor Activity, and T-cell Responses in a Dose-Ranging Phase I Trial of the Oncolytic Peptide LTX-315 in Patients with Solid Tumors. Clin Cancer Res. 2021 May 15;27(10):2755-2763. doi: 10.1158/1078-0432.CCR-20-3435. Epub 2021 Feb 4. PMID 33542073
- See also: Company webpage — http://www.lytixbiopharma.com